CLINICAL TRIAL: NCT05270850
Title: Clinical Study on Autologous Stromal Vascular Fraction(SVF) Treatment for Benign Airway Stenosis and Respiratory Tract Fistula
Brief Title: Clinical Study on Autologous Stromal Vascular Fraction(SVF) Treatment for Refractory Benign Airway Stenosis and Respiratory Tract Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of Department of Respiratory Medicine, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220210
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Benign Airway Stenosis; Respiratory Tract Fistula
Keywords: Stromal Vascular Fraction
MeSH Terms: conditions — Respiratory Tract Fistula | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional treatment for benign airway stenosis Including, but is not limited to laser, high-frequency electric knife, argon plasma coagulation (APC), cryotherapy, balloon dilation, and metal stent placement
  Interventions: Procedure: Control group
- SVF group (Experimental): SVF treatment following the conventional treatment for benign airway stenosis and respiratory tract fistula.
  Interventions: Procedure: SVF group

INTERVENTIONS:
Procedure: Control group — Conventional treatment for benign airway stenosis Including, but is not limited to laser, high-frequency electric knife, argon plasma coagulation (APC), cryotherapy, balloon dilation, and metal stent placement
  Arms: Control group
Procedure: SVF group — SVF treatment following the conventional treatment for benign airway stenosis and respiratory tract fistula
  Arms: SVF group

SUMMARY:
Benign airway stenosis and respiratory tract fistula are common types of airway injury. The diseases occurred after endogenous and exogenous stimuli (tuberculosis, tumor, surgery, tracheal intubation) causing damage to the airway mucosa, resulting in scar repair and irreversible loss of airway epithelium. Autologous adipose vascular fraction (stromal vascular fraction, SVF) is a mixture of cells obtained from adipose tissue through digestion and centrifugation, containing a variety of cell types, such as mesenchymal cells, endothelial progenitor cells, endothelial cells, pericytes, and macrophages. Previous studies have shown that SVF can achieve regeneration and wound healing through modulating the immune microenvironment, promoting angiogenesis, thereby promoting endogenous regeneration of the in situ adult stem cells. This project utilizes the tissue repair function of autologous SVF to treat benign airway stenosis and respiratory tract fistula. To clarify the efficacy and safety of autologous SVF in the treatment of airway injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 to 75
* Subjects diagnosed with benign airway stenosis, tracheoesophageal fistula(the sizes of the fistulas less than 2cm), and bronchopleural fistula
* Subjects willing to accept SVF treatment
* Subjects tolerant to the bronchoscope
* Subjects signed informed consent

Exclusion Criteria:

* Subjects with the following pulmonary diseases: asthma, active pulmonary tuberculosis, pulmonary embolism, pneumothorax, pulmonary hypertension, etc;
* Subjects with incomplete remission of malignant tumors or with incurable malignant tumors;
* Subjects with uncontrolled systemic infection;
* Subjects requiring anti-clotting drugs;
* Subjects with myocardial infarction, unstable angina, liver cirrhosis, acute glomerulonephritis, etc;
* Subjects with syphilis, HIV, HBV, HCV antibody positive;
* Subjects with Coagulation disorders such as hemophilia, giant platelet syndrome, thromboasthenia, etc;
* Subjects with severe renal damage, serum creatinine is more than 1.5 times the upper limit of the normal value;
* Subjects with liver disease or liver damage: ALT, AST, total bilirubin > 2 times the upper limit of the normal value;
* Subjects with a history of psychosis or suicide or epilepsy or other central nervous system diseases;
* Subjects with severe arrhythmias(e.g. ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or degree II above abnormal conduction;
* Subjects allergic to thrombin;
* Subjects accepted by any other clinical study within the first three months of the study;
* Subjects with poor compliance;
* Any other conditions might increase the risk of the patient or interfere with the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate for benign airway stenosis | within 3 months after administration
  The proportion of patients who is no need for endotracheal intervention and with stable clinical symptoms after SVF treatment
Cure rate for respiratory tract fistula | within 3 months after administration
  The proportion of patients who have complete closure of fistula, no need for endotracheal intervention and with stable clinical symptoms after SVF treatment

SECONDARY OUTCOMES:
Clinical complete remission time | within 3 months after administration
  The interval time of the first intratracheal interventional therapy needed again after SVF treatment
Times of unplanned treatment | within 3 months after administration
  The number of times a patient needs to be reviewed and treated by bronchoscopy
Incidence of complications associated with SVF treatment | within 3 months after administration
  Wound healing, sputum retention, etc. during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No